CLINICAL TRIAL: NCT06655116
Title: The Effect of Patient Education on Foot Care Behaviour and Diabetic Foot Self-Efficacy in Individuals With Type II Diabetes: A Randomised Controlled Study
Brief Title: Diabetic Foot Education
Status: Enrolling by invitation | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Hilal KAHRAMAN, Res. Asst. PhD, TC Erciyes University
Other Study IDs: 16.10.2024
Record Dates: First submitted 2024-10-16; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Diabetes Mellitus; Diabetic Foot Disease
Keywords: Diabetic Foot; Diabetes Mellitus; Patient Education
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Foot

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group
- Study Grup
  Interventions: Behavioral: Diabetic Foot Education

INTERVENTIONS:
Behavioral: Diabetic Foot Education — Patients in the intervention group will be interviewed and their diabetic foot knowledge will be evaluated. During the interview, the individual's knowledge about the definition of diabetic foot, risk factors, symptoms, treatment, complications, care and prevention will be evaluated.
  In order to systematically plan, implement and evaluate the training to be used in the intervention, it is aimed to implement androgogical training based on the 'Interpersonal Relations Theory'. In this context, the stages in the theory will be followed as follows.
  Groups: Study Grup

SUMMARY:
To determine the effect of foot care training given according to Interpersonal Relationship Theory on foot care behaviour and diabetic foot self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Diagnosis of Type 2 DM for at least 6 months,
* Not having received planned diabetic foot training before,
* Volunteering to participate in the study,

Exclusion Criteria:

* Neuropsychiatric drug use and disease that may affect education (Dementia- Alzheimer's and Mental Retardation etc.)
* Being visually impaired,
* Hearing impairment,
* Inability to speak Turkish,
* Presence of active diabetic foot ulcer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Erciyes University Health Application and Research Centre
Sampling Method: Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2024-10-26 (Estimated); Primary Completion 2024-11-26 (Estimated); Study Completion 2024-12-26 (Estimated)

PRIMARY OUTCOMES:
Descriptive Information Form: | 2 Minutes
  The descriptive information form, which was created by the researchers by reviewing the literature, consists of 16 items in total, including seven questions about individual characteristics (age, gender, height, weight, education level, family structure, smoking) and nine questions about the disease and diabetic foot (HbA1c value, number of years of living with diabetes, treatment(s) received, history of diabetic foot).
Diabetic Foot Self-Care Behaviour Scale | 5 minutes
  The Diabetic Outpatient Self-Care Behaviour Scale was developed by Yen-Fan Chin and Tzu-Ting Huang in 2013 (Chin & Huang, 2013). The Turkish validity and reliability study conducted by Bakır and Samancıoğlu Bağlama was published in 2021. The scale is a five-point Likert-type scale consisting of 7 items and two sections. The first part consists of four items including practices related to examining, washing and drying the soles of the feet and toes during the week. The three items in the second section are related to the use of shoes and lotion. The lowest score that can be obtained from the first section is 4 and the highest score is 20. The lowest score that can be obtained from the second section is 3 and the highest score is 15. The questionnaire is evaluated over the total score and the score that can be obtained varies between 7-35. As the score obtained from the scale increases, self-care behaviour increases.
Diabetic Foot Care Self-Efficacy Scale | 5 minutes
  The scale consisting of nine items is answered with an 11-digit visual scale ranging from 0-10. In the answers, the lowest value is expressed as 'I do not consider it sufficient at all' and the highest value is expressed as 'I consider it very sufficient'. The scale has no sub-dimensions and is evaluated on the total scale score. The lowest score that can be obtained from the scale is 0 and the highest score is 90. As the score obtained from the scale increases, the level of diabetic foot self-efficacy increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No